CLINICAL TRIAL: NCT01483378
Title: Increasing Use of the Vaccine Against Herpes Zoster/Shingles at NYULMC and Bellevue Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-02029
Record Dates: First submitted 2011-11-18; First posted 2011-12-01 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects who received the vaccine (Other): Patients in this arm were eligible for the herpes zoster vaccine and chose to receive it.
  Interventions: Other: Choosing to receive the vaccine
- Subjects who declined the vaccine (No Intervention)

INTERVENTIONS:
Other: Choosing to receive the vaccine
  Arms: Subjects who received the vaccine

SUMMARY:
The purpose of this study is to determine if vaccination rate of eligible patients at a major urban public hospital will increase by having ophthalmologists screen patients for eligibility and a nurse administer the vaccine in the General Eye Clinic.

DETAILED DESCRIPTION:
Patient vaccination behaviors will be assessed after 100 doses of the Zostavax vaccine are provided to underserved patients screened by ophthalmologists at the General Eye Clinic at a public hospital that does not normally provide the vaccine. A nurse will be at the clinic to administer the vaccine. Patients will be contacted by phone 1 month later and seen within 3 months in the Eye Clinic to determine whether there were any side effects.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Absence of evidence of immune compromise in the medical record
* Ability to speak and read English, Spanish or Chinese and give informed consent

Exclusion Criteria:

* Vulnerable patients, including the cognitively impaired, prisoners and employee
* FDA contraindications for Zostavax vaccine

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bellevue Hospital, New York, New York
  - NYU Langone Medical Center, New York, New York

REFERENCES:
- [Background] Ghaznawi N, Virdi A, Dayan A, Hammersmith KM, Rapuano CJ, Laibson PR, Cohen EJ. Herpes zoster ophthalmicus: comparison of disease in patients 60 years and older versus younger than 60 years. Ophthalmology. 2011 Nov;118(11):2242-50. doi: 10.1016/j.ophtha.2011.04.002. Epub 2011 Jul 23. PMID 21788078
- [Background] Hu AY, Strauss EC, Holland GN, Chan MF, Yu F, Margolis TP. Late varicella-zoster virus dendriform keratitis in patients with histories of herpes zoster ophthalmicus. Am J Ophthalmol. 2010 Feb;149(2):214-220.e3. doi: 10.1016/j.ajo.2009.08.030. Epub 2009 Nov 11. PMID 19909942
- [Background] Hurley LP, Lindley MC, Harpaz R, Stokley S, Daley MF, Crane LA, Dong F, Beaty BL, Tan L, Babbel C, Dickinson LM, Kempe A. Barriers to the use of herpes zoster vaccine. Ann Intern Med. 2010 May 4;152(9):555-60. doi: 10.7326/0003-4819-152-9-201005040-00005. PMID 20439573
- [Background] Lu PJ, Euler GL, Harpaz R. Herpes zoster vaccination among adults aged 60 years and older, in the U.S., 2008. Am J Prev Med. 2011 Feb;40(2):e1-6. doi: 10.1016/j.amepre.2010.10.012. PMID 21238856
- [Background] Oxman MN, Levin MJ, Johnson GR, Schmader KE, Straus SE, Gelb LD, Arbeit RD, Simberkoff MS, Gershon AA, Davis LE, Weinberg A, Boardman KD, Williams HM, Zhang JH, Peduzzi PN, Beisel CE, Morrison VA, Guatelli JC, Brooks PA, Kauffman CA, Pachucki CT, Neuzil KM, Betts RF, Wright PF, Griffin MR, Brunell P, Soto NE, Marques AR, Keay SK, Goodman RP, Cotton DJ, Gnann JW Jr, Loutit J, Holodniy M, Keitel WA, Crawford GE, Yeh SS, Lobo Z, Toney JF, Greenberg RN, Keller PM, Harbecke R, Hayward AR, Irwin MR, Kyriakides TC, Chan CY, Chan IS, Wang WW, Annunziato PW, Silber JL; Shingles Prevention Study Group. A vaccine to prevent herpes zoster and postherpetic neuralgia in older adults. N Engl J Med. 2005 Jun 2;352(22):2271-84. doi: 10.1056/NEJMoa051016. PMID 15930418
- [Background] Rimland D, Moanna A. Increasing incidence of herpes zoster among Veterans. Clin Infect Dis. 2010 Apr 1;50(7):1000-5. doi: 10.1086/651078. PMID 20178416
- [Background] Kaufman HE (ed) Herpes zoster ophthalmicus: preventing ocular complications through vaccination. Ophthalmology 2008; 115:S1-38
- [Derived] Jung JJ, Elkin ZP, Li X, Goldberg JD, Edell AR, Cohen MN, Chen KC, Perskin MH, Park L, Cohen EJ. Increasing use of the vaccine against zoster through recommendation and administration by ophthalmologists at a city hospital. Am J Ophthalmol. 2013 May;155(5):787-95. doi: 10.1016/j.ajo.2012.11.022. Epub 2013 Feb 6. PMID 23394910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We prospectively recruited eligible patients from the Bellevue Eye clinic until 100 patients were prescribed and received the vaccine. Recruitment occurred from January 9, 2012 to February 12, 2012.
Groups:
- Patients Who Received the Herpes Zoster Vaccine: These eligible subjects completed the survey and then chose to receive the herpes zoster vaccine for free.
- Patients Who Declined the Herpes Zoster Vaccine: These eligible subjects completed the survey and then declined to receive the herpes zoster vaccine for free.
Period: Overall Study
Arm/Group | Patients Who Received the Herpes Zoster Vaccine | Patients Who Declined the Herpes Zoster Vaccine
Started | 100 | 66
Completed | 100 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 170 patients were enrolled in the study, however 2 met FDA contraindications for herpes zoster vaccination and 2 already received the vaccine, so only 166 were included in the analysis.
Arm/Group | Survey Participants
Number analyzed (Participants) | 166
Age Continuous [Mean (Standard Deviation); unit: years]
  Age | 68 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 72
Region of Enrollment [Number; unit: participants]
  United States | 166

OUTCOME MEASURES:

1. Primary Outcome: Answers to Survey Questions
Description: All enrolled patients completed a survey of baseline characteristics, eligibility for the herpes zoster vaccine, and attitudes regarding herpes zoster vaccination. The survey results from patients who agreed to receive the herpes zoster vaccine were compared to the results of patients who declined to be vaccinated.
Time Frame: January 9, 2012 to February 12, 2012
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Groups:
- Patients Who Received the Herpes Zoster Vaccine: Patients who chose to receive the herpes zoster vaccine completed the survey. Primary outcomes reported are statistically significant answers to the survey questions.
- Patients Who Declined the Herpes Zoster Vaccine: Patients who declined to receive the herpes zoster vaccine completed the survey. Primary outcomes reported are statistically significant answers to the survey questions.
Arm/Group | Patients Who Received the Herpes Zoster Vaccine | Patients Who Declined the Herpes Zoster Vaccine
Number analyzed (Participants) | 100 | 66
Percentage of responders
  Subject reported receiving flu Vaccine last year | 89 [83 to 95] | 71.2 [60 to 82]
  Reported would receive the vaccine if recommended | 98 [95 to 100] | 74 [64 to 85]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were only collected and assessed for participants who received vaccine since there are no risks from the vaccine if the patient did not receive it.
Arm/Group | Subjects Who Received the Herpes Zoster Vaccine | Subjects Who Declined the Herpes Zoster Vaccine
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/0
Other Adverse Events (participants affected / at risk) | 11/100 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Who Received the Herpes Zoster Vaccine (N=100) | Subjects Who Declined the Herpes Zoster Vaccine (N=0)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less